CLINICAL TRIAL: NCT01112800
Title: Markers of Anthracycline-Related Cardiac Muscle Injury
Status: Withdrawn | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MARCI
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Osteosarcoma; Ewing's Sarcoma Family of Tumors; Rhabdomyosarcoma; Non-rhabdomyosarcoma Soft Tissue Sarcomas
Keywords: Anthracycline; Cardiac Muscle Injury; Doxorubicin; Doppler Imaging; Intermediate non-rhabdomyosarcoma soft tissue sarcomas; High-risk non-rhabdomyosarcoma soft tissue sarcomas
MeSH Terms: conditions — Osteosarcoma; Rhabdomyosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A blood sample will be collected at baseline, prior to and at the end of each doxorubicin infusion (48- or 72-hour) and following completion of chemotherapy for osteosarcoma, ESFT, rhabdomyosarcoma or intermediate and high-risk non-rhabdomyosarcoma soft tissue sarcomas.cTn-T and NT-BNP will be measured at baseline, prior to and at the end of each doxorubicin infusion (48- or 72-hour) and following completion of chemotherapy for osteosarcoma, ESFT, rhabdomyosarcoma or intermediate and high-risk non-rhabdomyosarcoma soft tissue sarcomas.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants: Previously untreated patients referred to St. Jude Children's Research Hospital (SJCRH) between the ages of 0 and 21 years with a diagnosis of osteosarcoma, ESFT, rhabdomyosarcoma and intermediate and high-risk non-rhabdomyosarcoma soft tissue sarcomas whose planned treatment includes administration of a cumulative anthracycline dose ≥ 375 mg/m2.

SUMMARY:
Anthracycline antibiotics are included in the chemotherapy regimens of approximately 82% of patients with bone cancer and 44% of those with soft tissue sarcoma diagnosed in childhood or adolescence. Impaired cardiac function occurs after treatment with anthracyclines. The frequency of impairment increases with increasing cumulative dose. There are inadequate data regarding the relationship between doxorubicin administration and changes in serum levels of cardiac troponin T (cTn-T) or I (cTn-I), N-terminal (NT) brain natriuretic peptide (BNP), or tissue Doppler imaging parameters.

This non-therapeutic study proposes a prospective, single arm study of serial changes in tissue Doppler imaging parameters, cTn-T and NT-BNP in children and adolescents with malignant bone and soft tissue tumors whose planned chemotherapy includes treatment with ≥ 375 mg/m2 of doxorubicin.

The proposed study will rigorously evaluate the usefulness of serial determinations of tissue Doppler imaging, cTn-T and NT-BNP for very early identification of anthracycline-related myocardial injury. Demonstration that one or more of these markers identifies subclinical myocardial damage and that biomarker or tissue Doppler imaging parameters exhibit a dose-response relationship with cumulative doxorubicin dose would facilitate intervention trials in patients at risk for anthracycline cardiomyopathy.

DETAILED DESCRIPTION:
The primary aim of this proposal is to serially evaluate imaging tests in previously untreated patients with osteosarcoma, Ewing's Sarcoma Family of Tumors(ESFT), rhabdomyosarcoma and intermediate and high-risk non-rhabdomyosarcoma soft tissue sarcomas whose planned treatment includes a cumulative doxorubicin dose ≥ 375 mg/m2 to determine if serial levels of one or more of these potential markers of cardiac muscle injury obtained prior to each infusion of doxorubicin and at the completion of chemotherapy correlate with increasing cumulative anthracycline exposure.

The secondary aim of the study is to estimate the proportion of patients with decreased (evaluation j - evaluation j+1) peak longitudinal systolic strain (ε) or strain rate (SR), peak radial systolic ε or SR, peak radial systolic myocardial velocity or peak longitudinal systolic myocardial velocity among those who have a shortening fraction (SF) ≥ 29% prior to each infusion of anthracycline. This study will evaluate whether the serum levels of cTn-T and/or NT-BNP will increase following doxorubicin administration. The study will evaluate whether the serum levels of cTn-T and/or NT-BNP will increase with increasing cumulative doxorubicin dose.

ELIGIBILITY:
Inclusion Criteria:

* Between 0 and 21 years of age
* Diagnosis of osteosarcoma, Ewing Sarcoma Family of Tumors, rhabdomyosarcoma, or intermediate or high-risk non-rhabdomyosarcoma soft tissue sarcoma
* Planned treatment includes administration of a cumulative anthracycline dose ≥ 375 mg/m2

Exclusion Criteria:

* Pregnant Females
* Patients with a history of cancer prior to the current malignancy
* Patients whose treatment will include radiation therapy to a volume that will include the heart

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Previously untreated patients referred to St. Jude Children's Research Hospital (SJCRH) between the ages of 0 and 21 years with a diagnosis of osteosarcoma, ESFT, rhabdomyosarcoma and intermediate and high-risk non-rhabdomyosarcoma soft tissue sarcomas whose planned treatment includes administration of a cumulative anthracycline dose ≥ 375 mg/m2.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Imaging measurement of potential cardiac muscle injury markers before and after cumulative anthracycline exposure. | 3 years
  This study will serially evaluate imaging tests in previously untreated patients with osteosarcoma, Ewing's sarcoma family of tumors, rhabdomyosarcoma and intermediate and high-risk non-rhabdomyosarcoma soft tissue sarcomas whose planned treatment includes a cumulative doxorubicin dose ≥ 375 mg/m2 to determine if serial levels of one or more of these potential markers of cardiac muscle injury obtained prior to each infusion of doxorubicin and at the completion of chemotherapy correlate with increasing cumulative anthracycline exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Green, MD, Principal Investigator — St. Jude Children's Research Hospital

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org